CLINICAL TRIAL: NCT06119373
Title: Initiation of Incremental Dialysis With Single Daily Icodextrin Exchange: a Randomized Controlled Trial
Brief Title: Incremental PD With Single Icodextrin Exchange
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wei Fang, Clinical Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-0224
Record Dates: First submitted 2023-10-13; First posted 2023-11-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Peritoneal Dialysis Complication; Residual Kidney Function; Survival; Health-related Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single daily icodextrin exchange group (Experimental): For incident peritoneal dialysis (PD) patients assigned to the experimental arm, PD is initiated with single daily exchange of 2-liter icodextrin-based dialysis solution. The daily dwell time ranges from 8-24 hours per day, depending on the patient's clinical conditions. Additional exchange(s) of glucose-based dialysis solution will be added to increase uremic toxins and fluid removal if necessary during the follow-up.
  Interventions: Other: Single daily icodextrin exchange
- Conventional PD group (Active Comparator): For incident peritoneal dialysis (PD) patients assigned to this arm, PD is initiated with 2 to 3 exchanges of 2-liter glucose-based solution. The daily dwell time ranges from 8-24 hours per day, depending on the patient's clinical conditions. Additional exchange(s) of glucose-based dialysis solution will be added to increase uremic toxins and fluid removal if necessary during the follow-up.
  Interventions: Other: Conventional PD group

INTERVENTIONS:
Other: Single daily icodextrin exchange — PD initiation with single daily exchange of 2-liter icodextrin-based dialysis solution.
  Arms: Single daily icodextrin exchange group
Other: Conventional PD group — PD is initiated with 2 to 3 exchanges of 2-liter glucose-based dialysis solution.
  Arms: Conventional PD group

SUMMARY:
Objectives: To investigate the efficacy and safety of single daily icodextrin exchange for initiation of incremental peritoneal dialysis (PD).

Subjects: Seventy-two incident PD patients.

Methods: A single-center randomized controlled trial.

Primary outcome: Change in residual kidney function in 48 weeks after recruitment.

DETAILED DESCRIPTION:
Incremental peritoneal dialysis (PD) has become a more prevalently adopted strategy in incident PD patients. There is significant variation in regimens of incremental PD. Initiation of PD with a single daily icodextrin exchange in patients with considerable residual kidney function is able to achieve successful water, sodium removal and solute clearance, while it has not been investigated and validated in randomized controlled trials.

This single-center, randomized, controlled study is to compare the effects of two prescriptions for initiation of incremental PD, a single daily icodextrin exchange versus 2-3 exchanges of glucose-based dialysate, on patients' residual kidney function, survival, peritonitis, and quality of life, in order to develop a new paradigm of incremental PD.

The primary outcome is change of residual kidney function, and the secondary outcomes include mortality, peritonitis-free survival, health-related quality of life, volume status, adequacy of small molecular solute clearance, and glucose exposure to dialysate.

Seventy-two eligible incident PD patients will be enrolled and randomly assigned to either the experimental or the control group in a ration of 1:1. Patients of the experimental group initiate PD with once daily exchange of 2-liter icodextrin dialysate, while those of the control group initiate PD with 2 to 3 exchanges of 2-liter glucose-based dialysate per day. All the enrolled patients will be prospectively followed up for 48 weeks. During the follow-up, the dose of dialysis would be incremental increased by adding exchange of glucose-based solution as required to accommodate for decline of RKF when at least one of the following indications is met: (1) clinical manifestations of uremia due to insufficient small solute clearance; (2) fluid overload which could not be corrected by salt and water intake restriction, increasing glucose concentration of dialysate, and administration of diuretics.

Residual kidney function, urine volume, peritoneal ultrafiltration, biochemical parameters, dialysate glucose exposure, volume status (measured by bioimpedence), and solute clearance are measured at baseline, and 24 and 48 weeks after recruitment, and are compared between groups. Quality of life is evaluated at baseline and 48 weeks by Kidney Disease Quality of Life-Short Form (KDQoL-SF) questionnaire, and are compared between two groups. Peritonitis rate for both groups are calculated and peritonitis-free survivals are compared. Differences in outcomes are evaluated by t test, Mann-Whitney test, or log-rank test where appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. male or female patients aged 18 to 75 years;
2. patients with chronic kidney disease stage 5 who are to start PD;
3. eGFR ≥ 5 ml/min;
4. urine output ≥ 800 ml/d.

Exclusion Criteria:

1. documented anaphylaxis with icodextrin or glucose-based dialysate;
2. concomitant severe chronic diseases such as malignancy, hepatitis, severe cardiac diseases, etc.;
3. ongoing severe infection;
4. planned or ongoing pregnancy or lactation;
5. currently enrolled in other clinical studies;
6. patients who have a life expectancy of <12 months;
7. refusal to give a written consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Residual kidney function | Up to 48 weeks after recruitment
  Change of residual kidney function in 48 weeks after PD initiation

SECONDARY OUTCOMES:
Mortality | Up to 48 weeks after recruitment
  The endpoint was death. The censored events include transfer to permanent hemodialysis, recovery of renal function, loss to follow-up, transfer to other dialysis centers, or to the end of study.
Peritonitis-free survival | Up to 48 weeks after recruitment
  The endpoint was first episode of PD-related peritonitis. The censored events were death, transfer to permanent hemodialysis, recovery of renal function, loss to follow-up, transfer to other dialysis centers, or to the end of study.
Health-related quality of life | Up to 48 weeks after recruitment
  Change of health-related quality of life assessed using Kidney Disease Quality of Life-Short Form in 48 weeks after recruitment. The form generates a score of 0 to 100, which represents better quality of life by a higher value.
Volume status | Up to 48 weeks after recruitment
  Change of volume status (Overhydration assessed by Bioelectric Impedance Analysis, etc.) in 48 weeks after recruitment
Adequacy of small molecular solute clearance | Up to 48 weeks after recuritment
  Change of weekly Kt/V and clearance of creatinine assessed using standard methods in 48 weeks after recruitment
glucose exposure to dialysate | Up to 48 weeks after recuritment
  change of glucose exposure to dialysate in 48 weeks after PD initiation

CONTACTS AND LOCATIONS:
Overall Officials: Wei Fang, MD., PhD., Principal Investigator — RenJi Hospital